CLINICAL TRIAL: NCT02251613
Title: Effectiveness of Olopatadine HCl Ophthalmic Solution, 0.1% Compared to Epinastine HCl Ophthalmic Solution, 0.05% in the Treatment of Allergic Conjunctivitis to Japanese Cedar Pollen
Brief Title: Effectiveness of Olopatadine HCl Ophthalmic Solution for the Treatment of Allergic Conjunctivitis in Japan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13-100-0009; UMIN000013943 (Registry Identifier: UMIN)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olopatadine (right or left, randomized) (Experimental): Olopatadine HCl ophthalmic solution, 0.1%, 1 drop in the right or left eye as randomized
  Interventions: Drug: Olopatadine HCl ophthalmic solution, 0.1%
- Epinastine (fellow eye) (Active Comparator): Epinastine HCl ophthalmic solution, 0.05%, 1 drop in the in the fellow eye
  Interventions: Drug: Epinastine HCl ophthalmic solution, 0.05%

INTERVENTIONS:
Drug: Olopatadine HCl ophthalmic solution, 0.1%
  Other Names: PATANOL®
  Arms: Olopatadine (right or left, randomized)
Drug: Epinastine HCl ophthalmic solution, 0.05%
  Arms: Epinastine (fellow eye)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Olopatadine Hydrochloride (HCl) ophthalmic solution 0.1% versus Epinastine HCl ophthalmic solution, 0.05% in a population of healthy, adult Japanese patients (20 years of age or older) with a history of allergic conjunctivitis to Japanese Cedar Pollen. Patients will be randomly assigned to receive Olopatadine HCl ophthalmic solution, 0.1% in one eye and Epinastine HCl ophthalmic solution, 0.05% in the fellow eye, after which a conjunctival allergy challenge (CAC) with Japanese cedar pollen will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Be Japanese and live in Japan;
* History of allergic conjunctivitis;
* Positive skin test reaction to Japanese cedar at Visit 1;
* Positive bilateral CAC reaction to the allergen at Visit 1 and Visit 2;
* Able and willing to avoid all disallowed medications during the specified period;
* Able to discontinue wearing contact lenses during the specified period;
* Sign Informed Consent;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History of hypersensitivity to the study drug or compounds;
* Any ocular condition that, in the opinion of the investigator, could affect the patient's safety;
* Ocular surgical intervention within 3 months or refractive surgery within 6 months prior to the start of the study;
* Presence of active ocular infection;
* Use of disallowed medications as specified in the protocol;
* Pregnant, nursing, or planning to become pregnant during the study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsunemitsu Senta, Study Director — Alcon Japan, Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study site located in Japan.
Pre-assignment Details: All subjects qualifying for treatment at Visit 3 were randomized. This reporting group includes all randomized participants (50).
Groups:
- Overall: Olopatadine HCl ophthalmic solution, 0.1%, and Epinastine HCl ophthalmic solution, 0.05%, administered contralaterally (1 drop in each eye), as randomized
Period: Overall Study
Arm/Group | Overall
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized participants.
Arm/Group | Overall
Number analyzed (Participants) | 50
Age, Customized [Number; unit: participants]
  20-29 years | 22
  30-39 years | 13
  40-49 years | 14
  ≥50 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Itching at 7 Minutes Post-CAC, Day 1
Description: A CAC (one drop of allergen solution to each eye) was performed 5 minutes after study medication instillation. Ocular itching was assessed by the patient for each eye at 7 (±1) minutes post-CAC and rated on a 0-4 scale (0=none, 4=incapacitating itch with irresistible urge to rub).
Time Frame: Day 1, 7 minutes post-CAC
Population: This analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Olopatadine 0.1%; Epinastine 0.05%: Ophthalmic solution, 1 drop instilled in 1 eye, as randomized.
Arm/Group | Olopatadine 0.1% | Epinastine 0.05%
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 50 | 50
units on a scale | 0.23 (0.31) | 0.37 (0.44)

2. Secondary Outcome: Mean Conjunctival Hyperemia at 20 Minutes Post-CAC, Day 1
Description: A CAC (one drop of allergen solution to each eye) was performed 5 minutes after study medication instillation. Conjunctival hyperemia (redness) was evaluated by the investigator based on biomicroscopy for each eye at 20 (±1) minutes post-CAC and rated on a 0-4 scale (0=none, 4=extremely severe).
Time Frame: Day 1, 20 minutes post-CAC
Population: This analysis population includes all randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Olopatadine 0.1% | Epinastine 0.05%
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 50 | 50
units on a scale | 0.89 (0.88) | 1.12 (0.95)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (December, 2013 - January, 2014). This analysis group includes all randomized subjects who received at least 1 dose of study medication.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered a study treatment regardless of whether or not the event has a causal relationship with the treatment, except for skin test and allergic symptom caused by CAC. AEs were obtained through solicited and spontaneous comments from the subjects.
Arm/Group | Olopatadine 0.1% | Epinastine 0.05%
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.